CLINICAL TRIAL: NCT03395106
Title: Developing and Evaluating Public Health Messages to Address Vaccine Hesitancy
Brief Title: Public Health Messages to Address Vaccine Hesitancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Immunization Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: H2016:390
Record Dates: First submitted 2017-12-12; First posted 2018-01-10 (Actual); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Vaccine Hesitancy
Keywords: vaccine; public health
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Intervention Model Description: Factorial design 2x2
Who Masked: Outcomes Assessor
Masking Description: Statisticians completing the analysis of the primary outcome will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Parent source + intuitive story content (Experimental)
  Interventions: Behavioral: Parent source; Behavioral: Intuitive content
- Doctor source + intuitive story content (Experimental)
  Interventions: Behavioral: Doctor source; Behavioral: Intuitive content
- Parent source + deliberative content (Experimental)
  Interventions: Behavioral: Parent source; Behavioral: Deliberative content
- Doctor source + deliberative content (Experimental)
  Interventions: Behavioral: Doctor source; Behavioral: Deliberative content

INTERVENTIONS:
Behavioral: Parent source — Having a parent feature prominently in a news story
  Arms: Parent source + deliberative content; Parent source + intuitive story content
Behavioral: Doctor source — Having a doctor feature prominently in a news story
  Arms: Doctor source + deliberative content; Doctor source + intuitive story content
Behavioral: Deliberative content — News story content includes process of weighing the risks/benefits of vaccinating, the importance of vaccines for community protection, and concludes with a recommendation to vaccinate.
  Arms: Doctor source + deliberative content; Parent source + deliberative content
Behavioral: Intuitive content — News story content focuses on the consequences of not vaccinating (including vaccine preventable diseases) and the decisional regret.
  Arms: Doctor source + intuitive story content; Parent source + intuitive story content

SUMMARY:
Views on vaccines range from those who are strongly supportive to those who are stridently opposed and will not budge from identity-based core beliefs about vaccines. In between these poles are numerous others who can delay, be reluctant (but still accept), or refuse/accept some vaccines for their children but not others. It is for these vaccine-hesitant parents that constitute the 'middle ground' of this spectrum where the most immediate and productive gains can be made towards enhancing vaccination acceptance and improving uptake. However, navigating this noisy communications environment is difficult, given the array of confusing and conflicting information available from multiple and competing sources. To date, there is no consensus on how best to use communication to respond to vaccine hesitancy. Building on two Canada-wide surveys of parents, the goal of this research is to identify which communication strategies show the greatest impact in reducing parental vaccine hesitancy and improving vaccination intentions.

The specific objectives are to:

1. Develop and pre-test four variations of news media stories that vary by source (parent versus physician) and content (intuitive versus deliberative);
2. Examine the impact of vaccine hesitant parents' exposure to vaccine communications that vary in source (parent versus physician) and content (intuitive versus deliberative) on primary (vaccine hesitant attitudes) and secondary (vaccine intentions) outcomes; and
3. Explore which media story variation may be more effective in improving vaccination attitudes and intentions for different parental decision-making styles (deliberative versus intuitive).

ELIGIBILITY:
Inclusion Criteria:

* Parents over 18 living in Canada with a YOUNGEST child is less than 24 months.

Exclusion Criteria:

* Parents who have a YOUNGEST child older than 24 months
* A parent who is pregnant, before the first trimester is complete

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 883 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-11-09 (Actual)

PRIMARY OUTCOMES:
Vaccine Hesitancy | Change in baseline measured up to 1 day after content delivery
  Parent Attitudes about Childhood Vaccines (PACV). The PACV is a validated 15 question survey on vaccine hesitancy.

SECONDARY OUTCOMES:
Intention to Vaccinate | Change in baseline measured up to 1 day after content delivery
  intention to vaccinate item using a 5 point likert scale ranging from very unlikely to vaccinate to very likely to vaccinate, and see if there is a one-response shift in participant intentions among vaccine hesitant parents.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Driedger, PhD, Principal Investigator — University of Manitoba
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pachur T, Spaar, M. Domain-specific preferences for intuition and deliberation in decision making. Journal of Applied Research in Memory and Cognition. 4:303-311, 2015.
- [Background] Opel DJ, Taylor JA, Zhou C, Catz S, Myaing M, Mangione-Smith R. The relationship between parent attitudes about childhood vaccines survey scores and future child immunization status: a validation study. JAMA Pediatr. 2013 Nov;167(11):1065-71. doi: 10.1001/jamapediatrics.2013.2483. PMID 24061681